CLINICAL TRIAL: NCT04313218
Title: Carbetocin Versus Misoprostol in Reducing Blood Loss During Cesarean Section in Low Risk Patients. A Retrospective Comparative Study
Brief Title: Carbetocin Versus Misoprostol. A Retrospective Comparative Study
Status: Completed | Type: Observational
Sponsor: Port Said University hospital (Other)
Responsible Party: Principal Investigator, waleed elsayed elrefaie, Assistant professor, Port Said University hospital
Other Study IDs: OBSGYN 1
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — carbetocin; Misoprostol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: recieved carbetocin 100ug iv after immediately after extraction of the fetus during cesarean section
  Interventions: Drug: Carbetocin
- B: women who received misoprostol 600ug rectally immediately before sterilization during cesarean section

INTERVENTIONS:
Drug: Carbetocin — iv infusion of 100ug carbetocin after extraction of the fetus during cesarean section
  Other Names: misoprostol
  Groups: A

SUMMARY:
Cesarean section is one of the most common surgeries practiced for save delivery of the fetus, however it is not a safe route of delivery its incidence is rising especially in high and middle income countries. The major concern is that the average blood loss during cesarean delivery is 487 ml, this amount is too close to the definition of postpartum hemorrhage by WHO as loss of 500 cc of blood in the first 24 hours after delivery making control of blood loss during cesarean delivery crucial to decrease maternal morbidities.This study aim to compare the use of misoprostol to carbetocin in reducing blood loss during cesarean section in low risk patients

DETAILED DESCRIPTION:
Cesarean section is one of the most common surgeries practiced for save delivery of the fetus, however it is not a safe route of delivery its incidence is rising especially in high and middle income countries. Although the WHO recommended cesarean section rate between 10 to 15% to decline the maternal mortality ratio and Neonatal mortality ratio, the incidence show sharp increase especially in Egypt to reach 52% of all deliveries. The major concern is that the average blood loss during cesarean delivery is 487 ml, this amount is too close to the definition of postpartum hemorrhage by WHO as loss of 500 cc of blood in the first 24 hours after delivery making control of blood loss during cesarean delivery crucial to decrease maternal morbidities. Many medications used to decrease blood loss especially placental site bleeding during cesarean section including oxytocin, ergometrine, synthetic prostaglandins and recently carbetocin.

Carbetocin is an oxytocin analogue containing eight amino acids .It binds to oxytocin receptors expressed on uterine muscles of pregnant women inducing tetanic uterine contractions for about 11 minutes after administration of 8-30ug intravenous followed by rhythmic uterine contractions that last for 60 to 120 minutes. Also it has a longer half life time than oxytocin and the recommended dose is 100ug IV.

Misoprostol is synthetic analogue to prostaglandin which is cheap heat stable uterotonic making it the alternative of choice to intravenous oxytocin in low resources countries. The recommended dose for prophylaxis against postpartum hemorrhage is 600μg while 800μg is used as a treatment.

In the lack of sufficient studies comparing the use of carbetocin to misoprostol to decrease blood loss during cesarean section we perform this study to compare the use of misoprostol to carbetocin in reducing blood loss during cesarean section.

Patients and Methods This was a retrospective comparative study conducted in Port Said General Hospital And Private practice in Port Said Egypt. Following approval of the study protocol by the ethical committee in Faculty of medicine Port Said University. The medical records of patients in the period from January 2018 to February 2019 were searched; women who underwent CS and were considered at low risk for postpartum including 1- singleton pregnancy, 2- less than previous four deliveries, 3- elective lower segment C.S, 4- C.S was done under general anesthesia 5- No medical disorders complicating pregnancy, 6- Placenta neither previa nor morbidly adherent, 7- Average amount of amniotic fluid, 8- No past history of postpartum hemorrhage and 9- No contraindications to Misopristol or Carbetocin 300 patients were eligible and were enrolled in this study. Women who received Carbetocin 100ug i.v (PABAL 100 micrograms/ml solution for injection, Ferring Pharmaceuticals Ltd) intra operative immediately after extraction of the fetus, were enrolled into group A and women who received misoprostol 600ug (cytotec 200ug tablet, Pfizer G.D. Searle LLC) rectally immediately before sterilization during caesarean section were enrolled into group B.

Maternal data (demographic and clinical), ultrasound findings, operative details, and postoperative characteristics were recorded in a database. The outcome measures of this study were the need for blood products transfusion, the amount of blood products transfusion, the operative time, operative complications uterine atony the need for surgical interventions to stop bleeding as uterine artery ligation and uterine compression sutures and the deficit in hemoglobin level.

ELIGIBILITY:
Inclusion Criteria:

* parity less than 4
* unscarred uterus or previous one cesarean section
* elective C.S
* general anesthesia

Exclusion Criteria:

* medical disorders complicating pregnancy
* more than one C.S
* selective C.S
* Risk factors for Postpartum hemorrhage

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: women who underwent CS and were considered at low risk for postpartum including 1- singleton pregnancy, 2- less than previous four deliveries, 3- elective lower segment C.S, 4- C.S was done under general anesthesia 5- No medical disorders complicating pregnancy, 6- Placenta neither previa nor morbidly adherent, 7- Average amount of amniotic fluid, 8- No past history of postpartum hemorrhage and 9- No contraindications to Misopristol or Carbetocin
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
blood loss | during operation
  reduction of blood loss during cesarean section operation

CONTACTS AND LOCATIONS:
Locations (1):
- Waleed Elsayed Elrefaie, Port Said, NY, Egypt

IPD SHARING:
Plan to Share IPD: No